CLINICAL TRIAL: NCT06190002
Title: Characteristics and Risk Factors for Invasive Fungal Infection in Hospitalized Patients With Acute-on-chronic Hepatitis B Liver Failure: A Retrospective Cohort Study From 2010 to 2023
Brief Title: Characteristics and Risk Factors for Invasive Fungal Infection With Acute-on-chronic Hepatitis B Liver Failure
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: KYLL-202310-035
Record Dates: First submitted 2023-12-17; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Acute-on-chronic Hepatitis B Liver Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- invasive fungal infection group and non-invasive fungal infection group: According to the presence or absence of invasive fungal infection, the patients were divided into invasive fungal infection group and non-invasive fungal infection group

SUMMARY:
This is a single-center retrospective study. The clinical data of patients with Acute-on-chronic Hepatitis B liver failure who were hospitalized in the Department of Hepatology, Qilu Hospital of Shandong University from January 2010 to July 2023 were collected.

DETAILED DESCRIPTION:
The clinical data of patients with Acute-on-chronic Hepatitis B liver failure who were hospitalized in the Department of Hepatology, Qilu Hospital of Shandong University from January 2010 to July 2023 were collected, including age, gender, HBsAg,HBeAg, serum hepatitis B virus DNA, alanine aminotransferase, aspartate aminotransferase, Platelet, white blood cell,neutrophilic granulocyte percentage, neutrophile granulocyte, total bilirubin, creatinine, international normalized ratio,procalcitonin,globulin. prothrombin time activity, 1, 3 - beta glucan D test, Galactomannan test, sputum culture, imaging CT and other indicators. Our study followed up patients with Acute-on-chronic Hepatitis B liver failure with fungal infection during hospitalization to clarify the clinical characteristics and risk factors of fungal infection in the development of Acute-on-chronic Hepatitis B liver failure , and to provide clinical prevention and treatment recommendations for fungal infection in patients with Acute-on-chronic Hepatitis B liver failure . Thus, the prognosis of patients can be improved and the survival rate can be increased.

ELIGIBILITY:
Inclusion Criteria:

* Acute liver function injury TBIL≥5mg/dl(85umol/L) and international normalized ratio (INR) ≥1.5 or PTA≤40% based on previously known chronic hepatitis B or compensated cirrhosis.
* Combined with ascites and/or hepatic encephalopathy within 4 weeks.
* HBsAg（+)>6 months

Exclusion Criteria:

* Patients died within 48 hours of admission or withdrew treatment.
* Combined with liver cancer and other extrahepatic organ malignant tumors, rheumatic diseases, hyperthyroidism.
* Age <18 years old.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The clinical data of patients with Acute-on-chronic hepatitis B liver failure hospitalized in the Department of Hepatology, Qilu Hospital of Shandong University from January 2010 to July 2023 were retrospectively collected. According to the inclusion criteria, 244 patients were finally included.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-01-20 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with invasive fungal infection | January 2010 to July 2023
  Invasive candidiasis: isolation of Candida in one or more blood cultures (candidemia) or from normal sterile body fluids. Candida colonization: Candida was isolated in non-sterile fluid without infection. Probable invasive aspergillosis: Detection of Aspergillus by direct examination and/or culture of respiratory specimens under imaging that is consistent with the presence of pulmonary infection. Probable invasive fungal infection(IFI) was defined as the presence of clinical features including lower respiratory tract mycosis (nodules, halo sign, air crescent sign, or cavity on chest CT scan) and a positive aspergillus culture in sputum specimen. In fact, the definitions of probable IFI and IFI are the same, except that probable IFI lacks mycological evidence.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chen Fan, MD,PhD, Study Chair — Qilu Hospital of Shandong University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Pauw B, Walsh TJ, Donnelly JP, Stevens DA, Edwards JE, Calandra T, Pappas PG, Maertens J, Lortholary O, Kauffman CA, Denning DW, Patterson TF, Maschmeyer G, Bille J, Dismukes WE, Herbrecht R, Hope WW, Kibbler CC, Kullberg BJ, Marr KA, Munoz P, Odds FC, Perfect JR, Restrepo A, Ruhnke M, Segal BH, Sobel JD, Sorrell TC, Viscoli C, Wingard JR, Zaoutis T, Bennett JE; European Organization for Research and Treatment of Cancer/Invasive Fungal Infections Cooperative Group; National Institute of Allergy and Infectious Diseases Mycoses Study Group (EORTC/MSG) Consensus Group. Revised definitions of invasive fungal disease from the European Organization for Research and Treatment of Cancer/Invasive Fungal Infections Cooperative Group and the National Institute of Allergy and Infectious Diseases Mycoses Study Group (EORTC/MSG) Consensus Group. Clin Infect Dis. 2008 Jun 15;46(12):1813-21. doi: 10.1086/588660. PMID 18462102